CLINICAL TRIAL: NCT07081477
Title: Effect of Ciprofol on Left Ventricular Outflow Tract Velocity-Time Integral in Elderly Patients Undergoing Painless Colonoscopy
Brief Title: Ciprofol's Influence on LVOT VTI in Elderly Painless Colonoscopy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY-20250307002-01
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Ciprofol
Keywords: Painless colonoscopy; Propofol; Left Ventricular Outflow Tract Velocity Time Integral
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- During anesthesia induction, ciprofol 0.2-0.5 mg/kg was intravenously injected (injection rate > 30s (Experimental): Group C
  Interventions: Drug: Intravenous Anesthetic Induction with Ciprofol for Painless Colonoscopy in Elderly Patients
- During anesthesia induction, propofol 1-2 mg/kg was intravenously injected (injection rate > 30s). (Active Comparator): Group P
  Interventions: Drug: Propofol Intravenous Anesthesia Induction for Painless Colonoscopy in Elderly Patients

INTERVENTIONS:
Drug: Intravenous Anesthetic Induction with Ciprofol for Painless Colonoscopy in Elderly Patients — Cirpropofol is a 2,6-disubstituted phenol derivative that introduces a cyclopropyl group based on the chemical structure of propofol, increasing its affinity with GABA receptors and stereoeffect, thus its effect is 4-5 times that of propofol. Studies have found that the incidence of hypotension, injection pain, and respiratory depression during cirpropofol anesthesia is lower than that of propofol.
  Arms: During anesthesia induction, ciprofol 0.2-0.5 mg/kg was intravenously injected (injection rate > 30s
Drug: Propofol Intravenous Anesthesia Induction for Painless Colonoscopy in Elderly Patients — Propofol has favorable pharmacokinetic properties with minimal residue. Currently, it is widely used for endoscopic procedure sedation, but there are still many limitations, such as a narrow therapeutic window, injection pain, hypotension, and respiratory depression.
  Arms: During anesthesia induction, propofol 1-2 mg/kg was intravenously injected (injection rate > 30s).

SUMMARY:
1. Objective:

   Primary: Compare the effect of Ciprofol vs Propofol on LVOT VTI at 2 minutes post-injection (T1) in elderly patients (≥65 years).

   Secondary: Assess hypotension incidence, injection pain, nausea/vomiting, hypoxia (SpO₂≤90%), bradycardia (HR<50 bpm), sedation success rate, induction/recovery times, procedure duration, drug doses, and patient satisfaction.
2. Design:

   Single-center, randomized, double-blind, controlled trial. Group C (Ciprofol):0.2-0.5 mg/kg IV induction (>30s injection). Group P (Propofol)::1-2 mg/kg IV induction (>30s injection). Rescue doses allowed (C: 0.1 mg/kg; P: 0.5 mg/kg; max 5 doses/15 min).
3. Participants:

   N = 120 elderly patients (65-80 years, ASA I-III, BMI 18-30 kg/m²) scheduled for elective painless colonoscopy.

   Exclusion: Significant cardiorespiratory, hepatic, renal, or neurological disorders; recent MI/unstable angina (≤6 months); NYHA ≥II; drug allergies; recent trial participation.
4. Key Assessments:

   Primary Endpoint: LVOT VTI (via transthoracic echocardiography, TTE) at T1.

   Secondary Endpoints:

   Adverse events (hypotension, pain, nausea/vomiting, hypoxia, bradycardia, body movement, awareness).

   Sedation success rate, induction/recovery times (MOAA/S scale), procedure time. Drug doses (induction, total, vasoactive agents). Patient satisfaction (5-point scale). LVEF and IVC Collapse Index (TTE at T0, T1, T2). Safety: Vital signs (HR, BP, SpO₂).
5. Statistical Analysis:

SPSS 26.0; α=0.05. Methods: t-test, RM-ANOVA, Mann-Whitney U, Chi-square/Fisher's exact, rank-sum tests.

This study aims to determine whether Ciprofol provides superior hemodynamic stability (as measured by LVOT VTI) and fewer adverse effects compared to Propofol for sedation in elderly patients undergoing painless colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA classification I-III;
2. Age ≥65 years and ≤80 years;
3. BMI between 18-30 kg/m2 (including the threshold);
4. Patients undergoing painless colonoscopy on an elective basis;
5. Subjects voluntarily participated in this study and signed an informed consent form.

Exclusion Criteria:

1. Those with respiratory depression or high risk of respiratory depression (e.g., sleep apnea syndrome, bronchial asthma, etc.);
2. Suffering from major diseases such as severe hepatic and renal insufficiency, neurological and psychiatric systems;
3. Suffering from severe arrhythmias such as severe aortic regurgitation, atrial fibrillation, tachycardia (heart rate > 120 beats/minute), atrioventricular block of degree II and above, myocardial infarction or unstable angina within 6 months before the examination, and NYHA classification grade II and above;
4. Allergy to or abuse of any medication used in the study;
5. Participation in another clinical trial within the last 3 months.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular outflow tract velocity time integral | Two minutes after administration
  The patient is in the left lateral position, using the same ultrasound equipment with standardized settings (gain, depth, frequency). Transthoracic Doppler echocardiography measurements are taken at the end of expiration.

SECONDARY OUTCOMES:
Left ventricular outflow tract velocity time integral | Perioperative
  The patient is in the left lateral position, using the same ultrasound equipment with standardized settings (gain, depth, frequency). Transthoracic Doppler echocardiography measurements are taken at the end of expiration.
Left ventricular ejection fraction | Perioperative
  The patient is in the left lateral position, using the same ultrasound equipment with standardized settings (gain, depth, frequency). Transthoracic Doppler echocardiography measurements are taken at the end of expiration.
Inferior Vena Cava Collapse Index | Perioperative
  Measure the maximum internal diameter (IVCmax) at end-expiration and minimum internal diameter (IVCmin) at end-inspiration of the inferior vena cava 1-2 cm from the right atrial entrance by ultrasound, and calculate according to the formula (IVCmax - IVCmin)/IVCmax × 100%.
adverse event | Perioperative
  The incidence of hypotension, injection pain, nausea, vomiting, hypoxemia (blood oxygen saturation ≤ 90%), bradycardia (heart rate < 50 beats per minute), body movement (unconscious limb movement of the patient), and intraoperative awareness.
Induction time | Perioperative
  Time from initial administration to Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≤1.
Procedure time | Perioperative
  The duration from colonoscopy insertion to withdrawal.
Awakening time | Perioperative
  The time from the end of the last administration to MOAA/S score equaling 5.
Induction drug dose , additional dose , total dose and vasoactive drug dose | Perioperative
Sedation success rate | Perioperative
  The number of patients who received up to 5 supplemental doses within 15 minutes after completing colonoscopy, without requiring rescue sedation, following the initial dose.
Patient satisfaction | Perioperative
  Patient satisfaction with anesthesia is divided into five options: very satisfied, satisfied, neutral, dissatisfied, and very dissatisfied.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT07081477/Prot_SAP_ICF_000.pdf